CLINICAL TRIAL: NCT04938947
Title: Effect of Resistance Training With Blood Flow Restriction on Motor Unit Hypertrophy in the Vastus Lateralis
Brief Title: Resistance Training and Blood Flow Restriction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Responsible Party: Principal Investigator, Tanner Reece, Graduate Teaching Assistant, University of Kansas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00147374
Record Dates: First submitted 2021-06-22; First posted 2021-06-25 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Blood Flow Restriction and Low-Intensity Resistance Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Intensity Resistance Training Group (Experimental): Participants in this group will complete 3 resistance training sessions per week for 6 weeks (18 sessions total). During each resistance training session, participants will perform 3 sets of bilateral leg-extensions (performed with both legs) to volitional failure (likely 8-12 repetitions) using 80% of their 1-repetition maximum (the most weight they are able to perform 1 complete repetition with, but not 2).
  Interventions: Other: High-Intensity Resistance Training
- Low-Intensity Resistance Training with Blood Flow Restriction Group (Experimental): Participants in this group will complete 3 resistance training sessions per week for 6 weeks (18 sessions total). During each training session, participants will perform 3 sets of bilateral leg-extensions (performed with both legs) to volitional failure using 30% of their 1-repetition maximum (the most weight they are able to perform 1 complete repetition with, but not 2). Participants in this group will perform all leg extensions with blood flow restriction cuffs applied to the proximal thigh of both legs. The pressure that the cuffs are inflated to will be calculated based on estimates of each subject's arterial occlusion pressure from their thigh circumference. Once the target pressure is reached, the cuffs will not be deflated until after the final set of the training session.
  Interventions: Device: Blood Flow Restriction Cuffs; Other: Low-Intensity Resistance Training

INTERVENTIONS:
Device: Blood Flow Restriction Cuffs — This intervention consists of inflatable cuffs that are designed to partially occlude veinous blood return from the lower extremities during resistance training.
  Other Names: Blood Flow Occlusion Cuffs
  Arms: Low-Intensity Resistance Training with Blood Flow Restriction Group
Other: Low-Intensity Resistance Training — This intervention consists of performing low-intensity bilateral (both legs at the same time) leg extensions using 30% of a participants 1 repetition maximum (the maximum weight an individual can complete 1 repetition with, but not 2) to volitional failure.
  Arms: Low-Intensity Resistance Training with Blood Flow Restriction Group
Other: High-Intensity Resistance Training — This intervention consists of performing high-intensity bilateral (both legs at the same time) leg extensions using 80% of a participants 1 repetition maximum (the maximum weight an individual can complete 1 repetition with, but not 2) to volitional failure.
  Arms: High-Intensity Resistance Training Group

SUMMARY:
The primary purposes of the proposed study is 1) To examine the changes of muscle fiber cross-sectional areas in the leg extensor muscles (vastus lateralis) pre- to post- 6 weeks of high-intensity resistance training and low-intensity resistance training with blood flow restriction and 2) To examine changes in motor unit size (a non-invasive measure of muscle fiber size) in the leg extensor muscles (vastus lateralis) pre- to post- 6 weeks of high-intensity resistance training and low-intensity resistance training with blood flow restriction.

DETAILED DESCRIPTION:
Specific Aims and Hypotheses:

Specific Aim 1: To examine the changes of type I and II (different types of muscle fibers) muscle fiber cross-sectional areas in the leg extensor muscles (vastus lateralis) pre- to post- 6 weeks of high-intensity resistance training and low-intensity resistance training with blood flow restriction. Hypothesis 1: Type I and II fiber cross-sectional area will increase following low-intensity resistance training with blood flow restriction, however, only cross-sectional area of type II fibers will increase post high-intensity resistance training.

Specific Aim 2: To examine changes in the size of the motor units that are active during low and high intensity contractions in the leg extensor muscles (vastus lateralis) pre- to post- 6 weeks of high-intensity resistance training and low-intensity resistance training with blood flow restriction. Hypothesis 2: The motor units that are active during low and high intensity contractions will increase in size from low-intensity resistance training with blood flow restriction, but only the motor units that are active during high intensity contractions will increase in size from high-intensity resistance training.

Specific Aim 3: To examine changes in whole muscle cross-sectional area as measured via ultrasound pre- to post- 6 weeks of high-intensity resistance training and low-intensity resistance training with blood flow restriction. Hypothesis 3: Whole muscle cross-sectional area will increase to similar degrees from both high-intensity resistance training and low-intensity resistance training with blood flow restriction.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Participants must not have participated in resistance training more than 5 times in the 6 months preceding the study.
* Participants must be healthy and free of any cardiovascular, metabolic or musculoskeletal conditions that may affect the results of the investigation.
* Participants must not have a history of severe hip, knee and/or ankle injuries, or any other pathological conditions that impair their motor control.
* Participants must not have any pre-existing cardiovascular conditions that involve blood flow/blood clotting.
* Participants who are currently taking blood thinners or any medications regulating blood pressures or heart rate will not be eligible to participate in the study.
* Female participants who are pregnant at the start of or who are planning to become pregnant during the resistance training intervention will not be eligible to participate in the study.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Determine changes in muscle fiber cross-sectional area | July 2021-May 2022
  A primary purpose of the study is to examine the changes of muscle fiber cross-sectional areas in the leg extensor muscles (vastus lateralis) pre- to post- 6 weeks of high-intensity resistance training and low-intensity resistance training with blood flow restriction
Determine changes in motor unit size | July 2021- May 2022
  Another primary purpose of the study is to examine changes in motor unit size (a non-invasive measure of muscle fiber size) in the leg extensor muscles (vastus lateralis) pre- to post- 6 weeks of high-intensity resistance training and low-intensity resistance training with blood flow restriction

CONTACTS AND LOCATIONS:
Locations (1):
- Robinson Center, Lawrence, Kansas, United States

IPD SHARING:
Plan to Share IPD: No